CLINICAL TRIAL: NCT01902004
Title: Treatment of Geriatric Depression With Mild Cognitive Impairment: A Double-blind Placebo-Controlled Trial of Namenda (Memantine) Augmentation of Lexapro (Escitalopram) in Depressed Patients at Least 60 Years of Age
Brief Title: Brain Aging and Treatment Response in Geriatric Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-01 MH097892; R01MH097892 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2013-07-17 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Mild Cognitive Impairment (MCI); Depression
Keywords: Major Depression; Geriatric Major Depression; Executive Cognitive Dysfunction; Mild Cognitive Impairment; Older Adults; Geriatric; Executive Cognitive Impairment; Quality of Life; Disability; Comorbidity; Medical Burden; Safety; Candidate Genes
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Depressive Disorder, Major | interventions — Escitalopram; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram and Memantine (Active Comparator): Participants will take a combination of Escitalopram and Memantine for 12 months
  Interventions: Drug: Escitalopram; Drug: Memantine
- Escitalopram and placebo (Active Comparator): Participants will take a combination of Escitalopram and placebo for 12 months
  Interventions: Drug: Escitalopram; Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — All subjects will receive 10 to 20mg of escitalopram open-label throughout the trial. Participants will begin taking one 10mg capsule once per day, and this dosage may be increased or decreased depending on the participant's response to the medication. Participants will continue on their assigned dosage of escitalopram until treatment completion.
  Other Names: Lexapro
Drug: Memantine — Memantine dosage will be 5 to 20mg a day. Participants will initially take one 5mg capsule once a day, which will be gradually increased to a maximum of 10mg capsules twice per day.
  Other Names: Namenda
  Arms: Escitalopram and Memantine
Drug: Placebo — Placebo pills will be taken in combination with the active Namenda (Memantine) pills. Participants will initially take 1 capsule per day, which will be increased to a maximum of 1 capsule twice per day.
  Other Names: inactive substance
  Arms: Escitalopram and placebo

SUMMARY:
The proposed project will evaluate the role of neuroimaging biomarkers of brain aging (i.e., neurodegenerative and vascular brain changes) and mild cognitive impairment in the patterns of treatment response to memantine combined with escitalopram compared to escitalopram and placebo.

DETAILED DESCRIPTION:
This study is designed to conduct a double-blind placebo-controlled trial of Namenda (Memantine) as an augmentation to Lexapro (Escitalopram) in depressed older adults 60 years of age and older. Throughout the course of the study, the investigators anticipate screening about 400 subjects to recruit 134 participants in the first four years. This study will require that the subjects complete up to 20 (twenty) visits in 12 (twelve) months to the study site during their participation. The purpose of this study is to determine whether Namenda (memantine) when taken in combination with Lexapro (escitalopram), may improve the quality of treatment response by making it faster and more complete, and also by improving thinking and memory in comparison to Lexapro taken with a placebo. Enrolled subjects will be provided with 10-20 mg of escitalopram for 12 months, and concurrently randomly assigned to either memantine or placebo groups. The investigators will also examine the safety and tolerability (how well the treatment works and the side effects) of a combination of Namenda and Lexapro as compared to placebo and Lexapro in subjects with major depressive disorder and mild cognitive impairment who are at least 60 years of age. Memantine is likely to accelerate and enhance antidepressant response to escitalopram and improve cognitive performance. Subjects with amnestic mild cognitive impairment or biomarkers of brain aging at baseline are likely to have preferential response to the combination of memantine and escitalopram compared to escitalopram and placebo, thus identifying a more personalized treatment approach in the high-risk subgroups for poor clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for major depressive disorder (recurrent and nonrecurrent course will be identified)
* Score of 16 or higher on the 24-item Hamilton Rating Scale for Depression (HDRS) at study entry
* Score of 24 or higher on the Mini-Mental State Exam (MMSE)
* Age 60 years old or older

Exclusion Criteria:

* History of psychiatric illness or a substance abuse disorder other than unipolar depression, diagnosed prior to the onset of the first depressive episode
* Presence of psychotic symptoms
* Severe or acute medical illness (e.g., major surgery, metastatic cancer, stroke, heart attack) 6 months prior to study entry
* Acute suicidal or violent behavior or history of suicide attempt within the year prior to study entry
* Presence of delirium, neurodegenerative dementia, Parkinson's disease, or any other central nervous system (CNS) diseases
* Toxic or metabolic abnormalities on laboratory examination
* Medications taken or medical illnesses present that could account for depression
* Active heart failure categorized as Class III or greater according to New York Heart Association criteria
* Heart attack or crescendo angina within the 3 months prior to study entry
* Symptomatic cardiac arrhythmias or symptomatic, hemodynamically significant mitral or aortic valvular disease
* Resting heart rate less than 50 beats per minute and a corrected QT (QTc) interval greater than 0.45 seconds
* Second or third degree atrioventricular block
* Systolic blood pressure greater than 180 mmHg or less than 90 mmHg and diastolic blood pressure greater than 105 mmHg or less than 50 mmHg at study entry
* Treated with depot neuroleptic therapy within 6 months prior to study entry
* Treated with any neuroleptic, antidepressant, anxiolytic medication (other than lorazepam), or over-the-counter CNS-active medications used for treatment of depression (e.g, St. John's Wort, kava-kava, melatonin) within 2 weeks (4 weeks for fluoxetine or monoamine-oxidase inhibitors [MAOIs]) prior to the first administration of study medication
* Known allergy to escitalopram or memantine or history of ineffective treatment with escitalopram or memantine for current depressive episode
* Requires concomitant therapy with any prescription or over-the-counter medications that have potentially dangerous interactions with either escitalopram or memantine
* Requires electroconvulsive therapy (ECT) or received ECT within 3 months prior to study entry
* Initiated psychotherapy within 3 months prior to study entry or will be initiating or terminating psychotherapy during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute - Neuropsychiatric Institute (NPI), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilpatrick LA, Krause-Sorio B, Siddarth P, Narr KL, Lavretsky H. Default mode network connectivity and treatment response in geriatric depression. Brain Behav. 2022 Apr;12(4):e2475. doi: 10.1002/brb3.2475. Epub 2022 Mar 1. PMID 35233974
- [Derived] Krause-Sorio B, Siddarth P, Kilpatrick L, Laird KT, Milillo MM, Ercoli L, Narr KL, Lavretsky H. Combined treatment with escitalopram and memantine increases gray matter volume and cortical thickness compared to escitalopram and placebo in a pilot study of geriatric depression. J Affect Disord. 2020 Sep 1;274:464-470. doi: 10.1016/j.jad.2020.05.092. Epub 2020 May 24. PMID 32663977
- [Derived] Grzenda A, Siddarth P, Laird KT, Yeargin J, Lavretsky H. Transcriptomic signatures of treatment response to the combination of escitalopram and memantine or placebo in late-life depression. Mol Psychiatry. 2021 Sep;26(9):5171-5179. doi: 10.1038/s41380-020-0752-2. Epub 2020 May 7. PMID 32382137
- [Derived] Lavretsky H, Laird KT, Krause-Sorio B, Heimberg BF, Yeargin J, Grzenda A, Wu P, Thana-Udom K, Ercoli LM, Siddarth P. A Randomized Double-Blind Placebo-Controlled Trial of Combined Escitalopram and Memantine for Older Adults With Major Depression and Subjective Memory Complaints. Am J Geriatr Psychiatry. 2020 Feb;28(2):178-190. doi: 10.1016/j.jagp.2019.08.011. Epub 2019 Aug 22. PMID 31519517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were excluded after being consented and prior to randomization. 5 were determined to be ineligible after completing the in-person screen visit in which they were consented. 15 withdrew consent before being randomized.
Period: Overall Study
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
Started | 48 | 47
Completed | 33 | 29
Not Completed | 15 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 8 | 22
  >=65 years | 34 | 39 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (6.9) | 72.8 (6.8) | 71.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 22 | 22 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 37 | 33 | 70
  African American | 4 | 2 | 6
  Hispanic | 3 | 8 | 11
  Other | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 95
Hamilton Depression Rating Scale Score [Mean (Standard Deviation); unit: units on a scale] — Clinician administered scale measures severity of depressive symptoms. This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
  units on a scale | 17.8 (2.3) | 17.7 (2.4) | 17.8 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale
Description: Clinician administered scale measures severity of depressive symptoms. This measure includes 24 items. Response options vary item to item and include the following ranges: [0-2], [0-3], and [0-4]. A score of 0 suggests absence of symptoms and/or difficulties and higher scores represent more severe difficulties. Possible overall score range [0-74], higher scores representing more severe difficulties.
Time Frame: Measured at 3 months; 6 months and 12 months
Population: The number of participants with available data at each time point differs due to participant dropout over the course of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
Number analyzed (Participants) | 48 | 47
units on a scale
  Baseline | 17.8 (2.3) | 17.7 (2.4)
  3 Months: number analyzed (Participants) | 35 | 32
  3 Months | 6.0 (4.5) | 6.7 (4.7)
  6 Months: number analyzed (Participants) | 33 | 29
  6 Months | 5.9 (5.2) | 6.9 (5.1)
  12 Months: number analyzed (Participants) | 23 | 21
  12 Months | 7.2 (5.8) | 5.4 (5.3)

2. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale
Description: Clinician administered item scale measures severity of depressive symptoms. The 10 items are measured on a 7-point scale ranging from 0 to 6; creating a total range of 0-60. A score of 0 suggests absence of symptoms and higher scores represent greater severity of depression.Severity gradations for the MADRS have been proposed (9-17 = mild, 18-34 = moderate, and ≥ 35 = severe). Treatment remission is defined as an endpoint total score ≤ 10.
Time Frame: Measured at 3 months; 6 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
Number analyzed (Participants) | 48 | 47
units on a scale
  Baseline | 16.7 (3.2) | 14.8 (3.5)
  3 Months: number analyzed (Participants) | 35 | 32
  3 Months | 7.1 (5.9) | 8.7 (5.5)
  6 Months: number analyzed (Participants) | 33 | 29
  6 Months | 6.0 (5.5) | 8.6 (4.5)
  12 Months: number analyzed (Participants) | 23 | 21
  12 Months | 8.8 (7.3) | 8.0 (6.5)

3. Secondary Outcome: Change in Cognitive Domain Scores
Description: Neuropsychological battery of tests which included the following domains: learning, delayed recall, and executive functioning. Raw scores were transformed to z-scores for each test score of interest for each participant, and then averaged. These z-scores were averaged within each neuropsychological domain to produce composite scores and then averaged over all tests to calculate a global performance score. Higher scores are indicative of better performance.
Time Frame: Measured at 6 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
Number analyzed (Participants) | 48 | 47
z score
  Baseline | .02 (.62) | -.04 (0.7)
  6 Months: number analyzed (Participants) | 33 | 29
  6 Months | 0.03 (.53) | -.1 (.67)
  12 Months: number analyzed (Participants) | 23 | 21
  12 Months | .15 (.67) | -.26 (.71)

4. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: The UKU (Udvalg for Kliniske Undersogelser) Side Effect Rating Scale organizes symptoms into 4 categories (i.e., Psychic, Neurologic, Autonomic, Other) containing 8-19 symptoms each. Each symptom receives a score for degree and causal relationship. Degree is scored between 0-3 with higher scores being more severe. Causal relationship is scored as improbable, possible, or probable.
Time Frame: Measured at 3, 6 months and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
Number analyzed (Participants) | 48 | 47
Participants
  3 Months: number analyzed (Participants) | 35 | 32
  3 Months | 3 | 2
  6 Months: number analyzed (Participants) | 33 | 29
  6 Months | 3 | 5
  12 Months: number analyzed (Participants) | 23 | 21
  12 Months | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Escitalopram and Memantine | Escitalopram and Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 41/48 | 41/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram and Memantine (N=48) | Escitalopram and Placebo (N=47)
Concentration Difficulties (Psychiatric disorders) | 4 | 5
Asthenia/Lassitude/Increased Fatigability (Psychiatric disorders) | 3 | 2
Sleepiness/Sedation (Psychiatric disorders) | 11 | 11
Failing Memory (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 0 | 1
Tension/Inner Unrest (Psychiatric disorders) | 4 | 3
Increased Duration of Sleep (Psychiatric disorders) | 1 | 3
Reduced Duration of Sleep (Psychiatric disorders) | 1 | 3
Increased Dream Activity (Psychiatric disorders) | 1 | 1
Accomodation Disturbance (Eye disorders) | 1 | 0
Increased Salivation (General disorders) | 0 | 1
Reduced Salivation (General disorders) | 4 | 7
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Micturtion Disturbances (Renal and urinary disorders) | 1 | 3
Polyuria/Polydipsia (Renal and urinary disorders) | 3 | 3
Orthostatic Dizziness (General disorders) | 3 | 4
Palpitations/Tachycardia (Cardiac disorders) | 0 | 1
Increased Tendancy to Sweating (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Weight Gain (Metabolism and nutrition disorders) | 1 | 2
Diminished Sexual Drive (Reproductive system and breast disorders) | 4 | 4
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 2
Ejaculatory Dysfunction (Reproductive system and breast disorders) | 1 | 1
Orgastic Dysfunction (Reproductive system and breast disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT01902004/Prot_SAP_000.pdf